CLINICAL TRIAL: NCT00617006
Title: Before and After Study Evaluating Deployment of the Sprixx GJ Personal Hand Hygiene Device in the Intra-Operative Environment
Brief Title: Potential Nosocomial Infection Prevention Via Modification of Anesthesia Intraoperative Aseptic Practice
Status: Completed | Type: Observational
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Harbor Medical Inc. (Industry)
Responsible Party: Matthew D. Koff M.D. M.S./Assistant Professor Anesthesiology and Critical Care Medicine, Dartmouth-Hitchcock Medical Center
Other Study IDs: CPHS# 20655
Record Dates: First submitted 2008-02-05; First posted 2008-02-15 (Estimated); Last update posted 2008-02-15 (Estimated); Status verified 2008-02

CONDITIONS: Nosocomial Infections
Keywords: Anesthesia Workspace; Hospital Acquired Infections; Hand Hygiene; Alcohol Based Cleanser; Bacterial Contamination
MeSH Terms: conditions — Cross Infection

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Environmental Bacterial Samples of Workspace
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Before (Control): Study group representative of standard practice
- After(Treatment): After treatment group with the personal hand hygiene device ie. Device Group.

SUMMARY:
We hypothesized that by improving hand hygiene compliance in the operative environment, we would reduce horizontal transmission of pathogenic bacteria to surgical patients.

DETAILED DESCRIPTION:
We performed an observational study evaluating provider adherence to these techniques. We then sought to increase hand hygiene compliance through the use of a point of care alcohol based hand hygiene device. We hypothesized that increased hand hygiene compliance would reduce bacterial contamination of the anesthesia workspace and peripheral intravenous tubing, and ultimately reducing overall morbidity and mortality secondary to a reduction in nosocomial infection rates.

ELIGIBILITY:
Inclusion Criteria:

* Patients present in operating rooms randomized to study.

Exclusion Criteria:

* Patients that were already enrolled in study and return to the operating room.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Operating Rooms were randomized and patients in these rooms were enrolled for the study.
Sampling Method: Probability Sample
Enrollment: 114 (Actual)
Dates: Start 2007-07; Primary Completion 2007-08 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
The presence of a positive culture on the previously sterile patient stopcock set, and the presence of multidrug resistant bacteria | Beginning and end of surgical case

SECONDARY OUTCOMES:
Reduction of bacterial contamination on predetermined sites on the anesthesia machine | Beginning and End of Surgical Case
Decreased length of stay | Postoperatively
Nosocomial infection rates | within 30 days postoperatively
Mortality | Within 30 days postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Matthew D Koff, M.D. M.S., Principal Investigator — Dartmouth-Hitchocck Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

REFERENCES:
- [Derived] Koff MD, Loftus RW, Burchman CC, Schwartzman JD, Read ME, Henry ES, Beach ML. Reduction in intraoperative bacterial contamination of peripheral intravenous tubing through the use of a novel device. Anesthesiology. 2009 May;110(5):978-85. doi: 10.1097/ALN.0b013e3181a06ec3. PMID 19352154